CLINICAL TRIAL: NCT02253368
Title: Home Sleep and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB14-0528
Record Dates: First submitted 2014-09-24; First posted 2014-10-01 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Overweight; Sleep
MeSH Terms: conditions — Overweight | interventions — Sleep

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Arm 1 (Active Comparator): Sleep Arm 1
  Interventions: Other: sleep
- Sleep Arm 2 (Active Comparator): Sleep Arm 2
  Interventions: Other: sleep

INTERVENTIONS:
Other: sleep

SUMMARY:
Bedtimes and wake-up times vary from person to person. The aim of this research is to examine the associations between sleep habits and metabolism in healthy people. In this study, the investigators will collect information on sleep-wake habits and how the body uses energy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-40 years
* Body mass index: 25.0 to 29.9 kg/m2
* Average habitual sleep duration of 6.5 hours or less per night (as confirmed by actigraphy)
* stable sleep habits for the past 6 months

Exclusion Criteria:

* obstructive sleep apnea or history of any other sleep disorder
* night or rotating shift work (current or in the past 2 years)
* habitual daytime naps
* recent (< 4 week) travel across time zones
* extreme chronotypes
* any acute or chronic medical condition
* diabetes
* prior or current eating or psychiatric disorders
* claustrophobia
* irregular menstrual periods, menopause, pregnancy,
* alcohol abuse, excessive caffeine intake, smoking, illegal drug use
* subjects who are currently following a weight loss regimen or any other special diet or exercise programs
* subjects who have received iv or oral contrast in the past 2 weeks
* use of any prescription medication that can affect sleep or metabolism with the exception of antihypertensive and lipid lowering agents as follows. Subjects who are taking anti-hypertensive medication and/or lipid-lowering agents will be included only if they are well controlled and on a stable regimen (no change in medications in the previous 3 months). However, beta-blockers and thiazide diuretics will not be allowed, as these medications are known to affect insulin sensitivity. Women will be required to not be on hormone replacement therapy.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in insulin sensitivity (SI) | The entire 4-week study is comprised of two 2-week periods: first 2-week period (baseline) and second 2-week period.
  Insulin sensitivity will be derived from minimal model analysis of mixed meal tolerance test. The mixed meal tolerance test is performed at the end of the first 2-week period and at the end of the second 2-week period. For each subject, the change from the first 2-week period in insulin sensitivity will be calculated.
Change from Baseline in total energy expenditure | The entire 4-week study is comprised of two 2-week periods: first 2-week period (baseline) and second 2-week period.
  Total energy expenditure will be derived from doubly labeled water method. For each subject, total energy expenditure will be calculated during each 2-week period and then the change from the first 2-week period in total energy expenditure will be calculated.
Change from Baseline in energy intake | The entire 4-week study is comprised of two 2-week periods: first 2-week period (baseline) and second 2-week period.
  Energy intake will be derived from doubly labeled water method and body composition analysis. For each subject, energy intake will be calculated during each 2-week period and then the change from the first 2-week period in energy intake will be calculated.
Change from Baseline in beta-cell function | The entire 4-week study is comprised of two 2-week periods: first 2-week period (baseline) and second 2-week period.
  Beta cell function will be derived from minimal model analysis of mixed meal tolerance test. The mixed meal tolerance test is performed at the end of the first 2-week period and at the end of the second 2-week period. For each subject, the change from the first 2-week period in beta-cell function will be calculated.
Change from Baseline in disposition index | The entire 4-week study is comprised of two 2-week periods: first 2-week period (baseline) and second 2-week period.
  Disposition index will be derived from minimal model analysis of mixed meal tolerance test. The mixed meal tolerance test is performed at the end of the first 2-week period and at the end of the second 2-week period. For each subject, the change from the first 2-week period in disposition index will be calculated.

SECONDARY OUTCOMES:
Change from Baseline in body weight | The entire 4-week study is comprised of two 2-week periods: first 2-week period (baseline) and second 2-week period.
  Weight will be derived from scale weight measurements. For each subject, their change in weight will be calculated during each period and then the change from the first 2-week period in body weight will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tasali, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Tasali E, Wroblewski K, Kahn E, Kilkus J, Schoeller DA. Effect of Sleep Extension on Objectively Assessed Energy Intake Among Adults With Overweight in Real-life Settings: A Randomized Clinical Trial. JAMA Intern Med. 2022 Apr 1;182(4):365-374. doi: 10.1001/jamainternmed.2021.8098. PMID 35129580

DOCUMENTS (1):
  • Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT02253368/ICF_000.pdf